CLINICAL TRIAL: NCT05855655
Title: Developing and Testing Internet-Based Mindfulness Intervention to Reduce Minority Stress and Promote HIV-Related Behavioral Health Among Young Adult Sexual Minority Men: Aim 3, A Randomized Controlled Trial
Brief Title: Developing an Online Mindfulness-based Intervention to Reduce Minority Stress and HIV Risk Among Young Adult MSM - Aim 3
Acronym: MBQR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2004002698-B; K23AT011173 (NIH)
Record Dates: First submitted 2023-05-04; First posted 2023-05-11 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Hiv; Minority Stress; Mental Health Wellness 1
Keywords: Mindfulness-based intervention; Sexual minority; LGBTQ; HIV prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The methodological approach includes a 2-arm trial of MBQR vs. a health education control group, with up to n=30 per arm (total Aim 3 sample size = up to 60 participants enrolled and randomized). The study is intended to evaluate the acceptability and feasibility of MBQR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Queer Resilience (MBQR) (Experimental): MBQR is an online, Zoom-based mindfulness course that meets 2.5 hour per week for ten weeks, facilitated by queer mindfulness teachers, with weekly home practice and additional reflection and reading activities that can be completed by participants independently via study website portal. In addition to the 10 weekly sessions there is an all-day retreat (6hrs) that takes place around week 6. The participants also meet one-on-one with the instructor(s) at the beginning and middle of class for a 30-minute welcome call and check in.
  Interventions: Behavioral: Mindfulness-Based Queer Resilience (MBQR)
- Health Education (Active Comparator): The online Health Education course is a self-paced program that can be largely completed independently (no group meeting, no all-day) by control group participants. The ten weekly modules are estimated to take around 30 to 90 minutes each to complete and consist of readings, videos, infographics, and other related activities (e.g., reflections, quizzes).
  Interventions: Behavioral: Mindfulness-Based Queer Resilience (MBQR)

INTERVENTIONS:
Behavioral: Mindfulness-Based Queer Resilience (MBQR) — This work aims to develop an internet-delivered MBI to address minority stress and its negative HIV-related health consequences experienced by young men who have sex with men (YMSM). This aim will examine the feasibility and acceptability of the internet-delivered mindfulness-based intervention (iMBI), called "Mindfulness-based Queer Resilience (MBQR)", for HIV prevention. The study will enroll and randomize a sample of 60 distressed, high-risk YMSM into one of two groups: MBQR intervention (n=30) or active control condition (n=30).

SUMMARY:
The overall aim of the research study is to develop and test a mindfulness-based program for young adult gay, bisexual, and queer men at risk for HIV (Brown University IRB approved protocol #2004002698). Researchers have completed Aims 1 and 2 of the broader study. Aim 1 used qualitative, community engaged methods, along with a quantitative online survey, to inform intervention development with the study population. Aim 2 involved seeking feedback on the developed mindfulness program through an open-pilot with 18 participants from the same study population (young adult gay, bisexual, and queer men at risk for HIV). The next phase of the intervention development (Aim 3 - registered here) will enroll and randomize a sample of 60 distressed, high-risk YMSM into one of two groups: MBQR intervention (n=30) or active control condition (n=30). Researchers aim to over-enroll YMSM of color (e.g., Black/Latinx YMSM) and anticipate the group to include approximately 50-60% Black/Latinx YMSM (or YMSM of color). Outcomes of feasibility and acceptability include rates of recruitment and retention, number of sessions attended, self-reported at-home practice of mindfulness, completion of assessment, and exit interviews.

DETAILED DESCRIPTION:
In 2017, gay, bisexual, and other men who have sex with men (MSM) made up 70% of new HIV infections in the U.S., and young adult MSM (age 18-34; YMSM) account for the majority of HIV cases. YMSM also experience prevalent, often co-occurring mental health issues, including depression, anxiety, and substance use, creating a "syndemic" condition surrounding HIV risk and suboptimal HIV testing.

A key driver of such disparities experienced by YMSM is minority stress. Experiences of identity-based discrimination lead to internalized stigma and maladaptive coping (e.g., emotion dysregulation, avoidant coping, impulsivity) The "downstream" effects of minority stress are poor mental health (depression and anxiety), increased sexual risk, and lack of engagement in key health services such as HIV testing due to anxiety related to identity disclosure to providers and anticipation of stigmatizing encounters. Recent evidence also suggests discrimination exposure is linked to heightened physiological stress response (cortisol level) that represents depletion of coping resources and increased risk for development of stress-linked psychological disorders (depression, anxiety). Therefore, reducing minority stress represents a promising transdiagnostic approach to reduce the burden of HIV and mental health issues experienced by YMSM.

Research suggests that Mindfulness-Based Interventions (MBIs) target mechanisms relevant to minority stress, including self-acceptance, emotional dysregulation, and avoidant coping. Therefore, as an individual-level intervention, MBIs may serve as an innovative HIV prevention intervention by lowering the syndemic risk among YMSM through reducing psychological symptoms, improving coping, and enhancing HIV-related behavioral health. However, no evidence-based MBIs have been tested for HIV prevention, and clinical and research evidence suggests further adaptation is warranted to improve its relevance and optimize engagement for YMSM.

This study aims to develop an internet-delivered MBI to address minority stress and its negative HIV-related health consequences experienced by YMSM. Specifically, the researchers propose to adapt, refine, and pilot-test an evidence-based MBI, Mindfulness-based Stress Reduction (MBSR), to promote mental and sexual health and HIV testing engagement among distressed, high-risk YMSM. Aims 1-3 will support the subsequent production and evaluation of the adapted intervention. To maximize reach, scalability, and availability to a population that experience challenges seeking in-person counseling and health services, the intervention will also be adapted for internet-based delivery.

Aim 1. (Previously Completed) Adapt MBSR for distressed, high-risk YMSM using internet delivery, guided by the ADAPT-ITT model. Researchers conducted iterative phases of formative research including online-based focus groups with YMSM, solicitation of feedback from stakeholders, and revision of intervention protocols. This process resulted in the first-draft of an internet-delivered, mindfulness-based intervention protocol for use with YMSM, known as "Mindfulness-Based Queer Resilience (MBQR)".

Aim 2. (Previously Completed - see ClinicalTrials.gov ID: NCT05540652) Refine intervention protocol by administering adapted materials to distressed, high-risk YMSM (n=18) through internet-based open pilot and gather feedback. Following integration of feedback, this process will result in a finalized protocol of an internet-delivered, mindfulness-based intervention protocol for YMSM.

Aim 3. (This is the focus of this Clinical Trial Registration) Examine the feasibility and acceptability of the internet-delivered mindfulness-based intervention (iMBI), called "Mindfulness-based Queer Resilience (MBQR)", for HIV prevention. Researchers will enroll and randomize a sample of 60 distressed, high-risk YMSM into one of two groups: MBQR intervention (n=30) or active control condition (n=30). They will aim to over-enroll YMSM of color (e.g., Black/Latinx YMSM) and anticipate the group to include approximately 50-60% Black/Latinx YMSM (or YMSM of color). The study will examine outcomes of feasibility and acceptability, such as rates of recruitment and retention, number of sessions attended, self-reported at-home practice of mindfulness, completion of assessment, and exit interviews.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male at birth,
* Being 18 to 34 of age,
* Identify as a cisgender man or nonbinary,
* Reside in the United States,
* Can read and speak English,
* Engaged in condomless anal sex with another man in past 6 months,
* Endorse distress, measured by the PHQ-9 and GAD-7,
* Possess a devise (phone, tablet, computer) that allows for online conferencing.
* HIV-negative at time of screening

Exclusion Criteria: Participants will be excluded from the study if they are determined to have symptoms that would prevent them from giving meaningful consent or participate in study activities including any of the following criteria:

* Significant cognitive impairment
* Psychosis
* Currently symptomatic and untreated bipolar disorder
* Imminent suicidal risk

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-04-08 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shufang Sun, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Following data collection, cleaning, and analysis, we plan to publish de-identified quantitative data at an open science data repository (e.g., Open Science Framework). De-identified qualitative data will be available upon request to the study PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Fall 2024

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-Based Queer Resilience (MBQR) | Health Education
Started | 34 | 34
Post-intervention Assessment | 34 | 33 (One participant from the control arm withdrew from the study)
6-month Follow-up | 30 (Four participants from the MBQR arm were lost-to-follow-up) | 33
Completed | 30 | 33
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Queer Resilience (MBQR) | Health Education | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.50 (4.12) | 27.15 (4.30) | 27.32 (4.18)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 31 | 60
  Gender Nonbinary, Nonconforming, Genderqueer | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 22 | 27 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Native American | 2 | 0 | 2
  Race: Asian | 3 | 5 | 8
  Race: Black | 5 | 4 | 9
  Race: Multiracial | 2 | 6 | 8
  Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Race: White | 16 | 14 | 30
  Race: Other | 6 | 5 | 11
Sexual Orientation [Count of Participants; unit: Participants]
  Gay | 26 | 26 | 52
  Straight | 0 | 0 | 0
  Bisexual | 1 | 1 | 2
  Pansexual | 4 | 1 | 5
  Other | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Online Mindfulness-Based Queer Resilience as Measured by Recruitment Rates
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Feasibility will be assessed via three measures. One measure of feasibility will be participant recruitment rates. The recruitment rate will be calculated by comparing the total number of participants screened eligible to those who were successfully enrolled in the study. See other primary outcomes for other measures used.
Time Frame: During recruitment period of study, up to 2 months
Population: Overall Number of Participants Analyzed represents number of participants eligible for study from the online screener.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-randomization: Number of participants under "Pre-randomization" represents numbers of individuals prior to randomization to either MBQR or control arms (e.g., number of individuals deemed eligible for study after screener).
Arm/Group | Pre-randomization
Number analyzed (Participants) | 223
Participants | 68

2. Primary Outcome: Feasibility of Online Mindfulness-Based Queer Resilience as Measured by Retention Rates: HIV/STI Testing Submission
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Feasibility will be assessed via three measures. One measure of feasibility will be participant retention rates, as measured by number of participants completing assessments. Data for one of the three assessments (i.e., HIV/STI testing submission) is reported here. Number of participants analyzed for each timepoint represent the number of participants who submitted any of the three assessments. See other primary outcomes for other measures used.
Time Frame: Baseline, Post-intervention (week 10), and 6-month Follow-up
Population: One participant from the control arm withdrew from the study between baseline and post-intervention assessments. Four participants from the MBQR arm were lost-to-follow-up at 6-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Queer Resilience (MBQR) | Health Education
Number analyzed (Participants) | 34 | 34
Participants
  Baseline: Completed all assessments | 34 | 34
  Post-intervention: number analyzed (Participants) | 34 | 33
  Post-intervention: Completed all assessments | 26 | 29
  6-month Follow-up: number analyzed (Participants) | 30 | 33
  6-month Follow-up: Completed all assessments | 27 | 28

3. Primary Outcome: Feasibility of Online Mindfulness-Based Queer Resilience as Measured by Retention Rates: Nail Sample Submission
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Feasibility will be assessed via three measures. One measure of feasibility will be participant retention rates, as measured by number of participants completing assessments. Data for one of the three assessments (i.e., nail sample submission for cortisol level testing) is reported here. Number of participants analyzed for each timepoint represent the number of participants who submitted any of the three assessments. See other primary outcomes for other measures used.
Time Frame: Baseline, Post-intervention (week 10), and 6-month Follow-up
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Queer Resilience (MBQR) | Health Education
Number analyzed (Participants) | 34 | 34
Participants
  Baseline | 30 | 28
  Post-intervention: number analyzed (Participants) | 34 | 33
  Post-intervention | 23 | 26
  6-month Follow-up: number analyzed (Participants) | 30 | 33
  6-month Follow-up | 23 | 24

4. Primary Outcome: Feasibility of Online Mindfulness-Based Queer Resilience as Measured by Retention Rates: Survey Submission
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Feasibility will be assessed via three measures. One measure of feasibility will be participant retention rates, as measured by number of participants completing assessments. Data for one of the three assessments (i.e., post-intervention and 6-month follow-up survey submission) are reported here. Number of participants analyzed for each timepoint represent the number of participants who submitted any of the three assessments. See other primary outcomes for other measures used.
Time Frame: Baseline, Post-intervention (week 10), and 6-month Follow-up
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Queer Resilience (MBQR) | Health Education
Number analyzed (Participants) | 34 | 34
Participants
  Baseline | 34 | 34
  Post-intervention: number analyzed (Participants) | 34 | 33
  Post-intervention | 33 | 31
  6-month Follow-up: number analyzed (Participants) | 30 | 33
  6-month Follow-up | 28 | 32

5. Primary Outcome: Feasibility of Online Mindfulness-Based Queer Resilience as Measured by Engagement
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Feasibility will be assessed via three measures. One measure of feasibility will be engagement with the MBQR program (i.e, adherence to the prescribed intervention), which will be assessed by class attendance data. The average number of sessions that participants attended the MBQR sessions is reported here.
Time Frame: During intervention period (10 weeks)
Population: The health education program was hosted on a website and did not include weekly sessions; therefore, class attendance data are not applicable, and no data were collected for that arm.
Measure: Mean (Standard Deviation); unit: Sessions
Arm/Group | Mindfulness-Based Queer Resilience (MBQR) | Health Education
Number analyzed (Participants) | 34 | 0
Sessions | 7.18 (3.43) |

6. Primary Outcome: Acceptability of Online Mindfulness-Based Queer Resilience as Measured by the Client Satisfaction Questionnaire
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Acceptability will be assessed using three measures. One such measure of acceptability will be via acceptability ratings using the validated 8-item Client Satisfaction Questionnaire (CSQ-8). Participants rated each item on a four-point Likert scale. Total scores for the CSQ-8 range from 8 to 32, with higher values indicating higher satisfaction. See other primary outcomes for other measures used.
Time Frame: Post-intervention (week 10)
Population: One participant from the control arm withdrew from the study during intervention period (i.e., before post-intervention assessments) and did not complete the post-intervention assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mindfulness-Based Queer Resilience (MBQR) | Health Education
Number analyzed (Participants) | 34 | 33
Scores on a scale | 26.61 (3.60) | 18.25 (5.47)

7. Primary Outcome: Acceptability of Online Mindfulness-Based Queer Resilience as Measured by a Session Evaluation Form
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Acceptability will be assessed using three measures. One such measure of acceptability will be via a session evaluation form that provides both qualitative and quantitative feedback on the study intervention using 10 questions, rated on a four-point Likert scale, and 6 free response questions. The quantitative data is reported here. Total scores range from 10 to 40, with higher values indicating higher satisfaction. See other primary outcomes for other measures used.
Time Frame: Post-intervention (week 10)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mindfulness-Based Queer Resilience (MBQR) | Health Education
Number analyzed (Participants) | 34 | 33
Scores on a scale | 33.27 (4.89) | 26.22 (5.92)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 6 months
Arm/Group | Mindfulness-Based Queer Resilience (MBQR) | Health Education
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT05855655/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT05855655/SAP_001.pdf
  • Informed Consent Form (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT05855655/ICF_002.pdf